Modification and evaluation of the DECIDE intervention to improve parentprovider interactions in low-income parents of adolescents with Disruptive Impulse Control, and Conduct Disorders

NCT number: NCT04445155

Date: 12/13/2023

Statistical Analysis Plan for the DECIDE Parent-Provider Intervention Study

The statistical analysis plan was changed from the original statistical analysis plan in the protocol because the study design was changed. Originally, there was a control group planned (treatment as usual); Instead, the study design was changed to a pre/post design, with outcomes collected pre- and post-intervention for three sample populations: 1) Providers; 2) Parents; and 3) a second group of providers (referred to as Provider Substudy).

SAS version 9.4 (Cary, NC) was used for statistical analysis. The alpha level was set at 0.05 for all statistical tests. For each outcome, change scores were calculated as post-intervention score minus pre-intervention score. Next, the change scores were tested for normality using the Shapiro-Wilk test. If the If the change scores were not normally distributed, then a Wilcoxon signed-rank test was conducted to see if the distribution of the outcome data was different from pre- to post-intervention. If the change scores were normally distributed, then a paired t-test was conducted to test whether the mean difference was not equal to zero. As pre- and post-intervention outcome data was available for only 3 parents, there were no statistical analyses conducted with the parent outcome data; thus, statistical tests were only generated for the Provider and Provider Subgroup outcomes.